CLINICAL TRIAL: NCT00405730
Title: Nepafenac 0.1% Eye Drops, Suspension Compared to Ketorolac Trometamol 0.5% Eye Drops, Solution and Placebo (Nepafenac Vehicle) for the Prevention and Treatment of Ocular Inflammation and Ocular Pain Associated With Cataract Surgery: European Study
Brief Title: Nepafenac 0.1% Eye Drops, Suspension Compared to Ketorolac Trometamol 0.5% Eye Drops, Solution and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-65; 2005-002647-35
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-04

CONDITIONS: Cataracts
Keywords: Cataracts
MeSH Terms: conditions — Cataract | interventions — nepafenac; Ophthalmic Solutions; Suspensions; Ketorolac; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nepafenac (Experimental): One drop in the study eye 3 times daily for 23 days
  Interventions: Drug: Nepafenac 1mg/ml eye drops, suspension
- Ketorolac Trometamol (Active Comparator): One drop in the study eye 3 times daily for 23 days
  Interventions: Drug: Ketorolac Trometamol 5 mg/ml eye drops, solution
- Nepafenac Vehicle (Placebo Comparator): One drop in the study eye 3 times daily for 23 days
  Interventions: Other: Nepafenac vehicle eye drops

INTERVENTIONS:
Drug: Nepafenac 1mg/ml eye drops, suspension — One drop in the study eye 3 times daily for 23 days
  Arms: Nepafenac
Drug: Ketorolac Trometamol 5 mg/ml eye drops, solution — One drop in the study eye 3 times daily for 23 days
  Arms: Ketorolac Trometamol
Other: Nepafenac vehicle eye drops — One drop in the study eye 3 times daily for 23 days
  Arms: Nepafenac Vehicle

SUMMARY:
To evaluate the safety and efficacy of Nepafenac 1 mg/ml Eye Drops, Suspension, compared to Placebo and Ketorolac Trometamol 5 mg/ml Eye Drops, Solution for the prevention and treatment of ocular inflammation and ocular pain after cataract extraction with IOL implantation

ELIGIBILITY:
Inclusion Criteria:

* Patients (18 years or older) of any race and either sex, requiring cataract extraction with planned implantation of a posterior chamber intraocular lens.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 18.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with Day 14 Cure | Day 14
  Cure is defined as aqueous cells score = 0 and aqueous cells score = 0 at Day 14.

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux, Bordeaux, France

REFERENCES:
- [Result] Nardi M, Lobo C, Bereczki A, Cano J, Zagato E, Potts S, Sullins G, Notivol R. Analgesic and anti-inflammatory effectiveness of nepafenac 0.1% for cataract surgery. Clin Ophthalmol. 2007 Dec;1(4):527-33. PMID 19668532